CLINICAL TRIAL: NCT03904381
Title: Efficacy and Safety of XEN® Gel Stent and Post-operative Management in Patients With Open Angle Glaucoma Compared to Classic Glaucoma Surgeries (Trabeculectomy and Sclerectomy) as Well as Other Minilally Invasive Glaucoma Surgery (MIGS)
Brief Title: Efficacy and Safety of XEN® Gel Stent and Post-operative Management in Patients With Open Angle Glaucoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wroclaw Medical University (Other)
Collaborators: Wrocław University of Science and Technology (Other)
Responsible Party: Principal Investigator, Joanna Przeździecka-Dołyk, Investigator, Wroclaw Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STM.C240.17.037
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Open-angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- stand-alone procedure of XEN implantation in phakic eyes (Active Comparator)
  Interventions: Drug: 5-fluorouracil; Procedure: Transconjunctival needling; Procedure: Transconjunctival revision
- stand-alone procedure of XEN implantation in pseudophakic eyes (Active Comparator)
  Interventions: Drug: 5-fluorouracil; Procedure: Transconjunctival needling; Procedure: Transconjunctival revision
- XEN implantation combined with cataract extraction (Active Comparator)
  Interventions: Drug: 5-fluorouracil; Procedure: Transconjunctival needling; Procedure: Transconjunctival revision

INTERVENTIONS:
Drug: 5-fluorouracil — 5-fluorouracil subconjunctival injections were a first-choice therapy for bleb failure and were administered according to predetermined criteria.
Procedure: Transconjunctival needling — Transconjunctival needling was administered according to predetermined criteria.
Procedure: Transconjunctival revision — Transconjunctival revision was administered according to predetermined criteria.

SUMMARY:
To evaluate the efficacy of postoperative management with 5-fluorouracil injections after XEN Gel Stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of primary open angle glaucoma
* trabecular meshwork visible in gonioscopy
* medicated IOP of ≥ 15 mmHg and ≤ 35 mmHg
* taking 1 to 5 IOP-lowering medications
* area of healthy, free and mobile conjunctiva in the target quadrant (superior-nasal)
* signed inform consent

Exclusion Criteria:

* angle closure glaucoma
* secondary open angle glaucoma
* previous glaucoma shunt/valve in the target quadrant
* presence of conjunctival scarring, prior conjunctival surgery or other conjunctival pathologies (e.g., pterygium) in the target quadrant
* active inflammation (e.g., blepharitis, conjunctivitis, keratitis, uveitis)
* active iris neovascularization or neovascularization of the iris within 6 months of the surgical date
* anterior chamber intraocular lens
* presence of intraocular silicone oil
* vitreous present in the anterior chamber
* impaired episcleral venous drainage (e.g., Sturge-Weber or nanophthalmos or other evidence of elevated venous pressure)
* known or suspected allergy or sensitivity to drugs required for the surgical procedure or any of the device components (e.g., porcine products or glutaraldehyde)
* history of dermatologic keloid formation
* previous photorefractive keratectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Unqualified success | 5 years
  Unqualified success of glaucoma treatment, defined as a postoperative IOP <18 mmHg and >20% reduction compared with the baseline value, achieved without use of any antiglaucoma medication and with no detected glaucoma progression as assessed at the final follow-up visit.

SECONDARY OUTCOMES:
Qualified success score A | 5 years
  Qualified success of glaucoma treatment, defined as a postoperative IOP <21 mmHg and >20% reduction compared with the baseline value, achieved with or without use of antiglaucoma medication and with no detected glaucoma progression as assessed at the final follow-up visit.
Qualified success score B | 5 years
  Qualified success of glaucoma treatment, defined as a postoperative IOP < 18 mmHg and >20% reduction compared with the baseline value, achieved with or without use of antiglaucoma medication and with no detected glaucoma progression as assessed at the final follow-up visit.
Qualified success score C | 5 years
  Qualified success of glaucoma treatment, defined as a postoperative IOP ≤15 mmHg and >40% reduction compared with the baseline value, achieved with or without use of antiglaucoma medication and with no detected glaucoma progression as assessed at the final follow-up visit.

OTHER OUTCOMES:
Glaucoma Progression | 5 years
  Glaucoma progression was evaluated with the Hodapp-Parrish-Anderson Glaucoma Grading Scale (GGS).
  Staging according to the standards given in bibliography (Budenz et all in 2002)
Change in thickness of the retinal nerve fiber layer (RNFL) | 5 years
  Difference in thickness of the retinal nerve fiber layer during the observation time frame.
Change in thickness of ganglion cell complex (GCC) | 5 years
  Difference in thickness of ganglion cell complex during the observation time frame.
Short term changes in IOP after surgery | 5 years
  Evaluated with the use of water drinking test.
Refractive error | 5 years
  Change in refractive error after glaucoma procedures
Best-corrected visual acuity | 5 years
  Evaluated on the fixed charts by trained optometrist
Visual field (VF) | 5 years
  Detection of the visual field abnormalities on the standard machine and during screening procedures
Disc damage likelihood scale (DDLS) | 5 years
  Evaluation disc damage likelihood scale based on the fundus photographs
Peripapillar and macular vessels density | 5 years
  Measured on the custom-derived protocol and manufacturer software macular and peripapillar vessels density - Angio OCT (OCTA)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Misiuk-Hojło, Professor, Study Chair — Medical University of Wrocław; Ewa Wałek, Principal Investigator — Medical University of Wrocław
Locations (1):
- Department of Ophthalmology, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Budenz DL, Rhee P, Feuer WJ, McSoley J, Johnson CA, Anderson DR. Comparison of glaucomatous visual field defects using standard full threshold and Swedish interactive threshold algorithms. Arch Ophthalmol. 2002 Sep;120(9):1136-41. doi: 10.1001/archopht.120.9.1136. PMID 12215086
- [Background] Susanna R Jr, Vessani RM. Staging glaucoma patient: why and how? Open Ophthalmol J. 2009 Sep 17;3:59-64. doi: 10.2174/1874364100903020059. PMID 19834563